# 知情同意书

项目名称: 嵌合抗原受体 T 细胞免疫疗法(CAR-T)治疗难治性膜

性肾病的安全性和有效性研究

研究单位: 空军军医大学第一附属医院(西京医院)肾脏内科

主要研究者: 何丽洁

研究年限: 2025年08月01日-2028年07月31日

版本号: <u>V3.0</u>

版本日期: 2025年10月10日

尊敬的患者:

您将被邀请参加一项"单中心前瞻性探索性临床试验"的试验。该研究由何丽洁 副教授负责。本次研究将严格遵从《赫尔辛基宣言》和我国相关的法律法规要求。

在您决定是否参加该项临床研究之前,请仔细阅读以下内容,它可以帮助您 充分了解为何要进行该项研究、研究的程序和期限、参加研究后可能给您带来的 益处、风险和不适。您可以和您的亲属、朋友一起讨论,询问负责研究的医生, 他/她将为您解释您对于此研究的任何疑问,帮助您做出最终决定。

#### 一、研究背景

本研究是一项探索嵌合抗原受体 T 细胞免疫疗法(CAR-T)治疗难治性膜性 肾病的安全性和有效性的临床研究。以下是为您提供的研究背景信息,希望能帮 助您理解本研究的意义。

膜性肾病是一种常见的自身免疫性肾脏疾病,其根本原因是体内的免疫系统(主要是 B 细胞)产生了攻击肾脏的"自身抗体",导致肾脏损伤和严重的蛋白尿。目前,针对这种疾病的一线治疗,如钙调磷酸酶抑制剂、环磷酰胺、利妥昔单抗等免疫抑制药物均旨在清除产生抗体的 B 细胞。然而,约有三分之一的患者对现有治疗反应不佳,成为"难治性"患者,面临肾功能恶化的风险。因此,我们需要为这部分患者寻找新的治疗方案。

CAR-T 疗法是一种新型的精准免疫治疗方法。它的基本原理是从患者血液中提取自身的 T 细胞,在体外通过基因工程技术进行改造,使其能够精准识别并清除体内特定的异常细胞,如产生有害抗体的 B 细胞,然后将这些改造后的细胞回输到患者体内。这种疗法的一个重要潜在优势是,回输的细胞可能在体内长期存活,从而实现一次治疗、长期有效的可能。

近年来,CAR-T 疗法在肿瘤治疗中取得成功后,也开始应用于自身免疫性疾病领域。初步研究表明,它在治疗系统性红斑狼疮等自身免疫病中取得了令人鼓舞的疗效,且安全性总体可控,最常见的不良反应是通常为轻至中度的"细胞因子释放综合征"。

鉴于膜性肾病同样是由 B 细胞介导的自身免疫病,我们推测 CAR-T 疗法也可能为难治性膜性肾病患者带来希望。因此,我们计划开展本研究,旨在初步评估 CAR-T 疗法用于治疗难治性膜性肾病的安全性与有效性。

### 二、研究目的

当前,难治性膜性肾病患者对于一线免疫或靶向治疗无应答,进展为终末期肾脏病的风险显著增高。因此,仍需进一步探索难治性膜性肾病的有效治疗手段。 CAR-T细胞在自身免疫性疾病临床研究中的成果提示其在难治性膜性肾病中可能具有较好的潜力与应用前景。因此,我们的研究目的是通过前瞻性、小样本临床试验初步探索 CAR-T 疗法在难治性膜性肾病中的安全性及有效性,以期为难治性膜性肾病提供更好的治疗策略。

#### 三、研究设计

本研究是一项由西京医院肾脏内科何丽洁副教授团队发起的为单中心小样本探索性试验。

您将在接受标准对症和支持疗法的基础上,接受单次自体 CD19 CAR-T 细胞治疗。您在接受 CAR-T 细胞治疗前 1-4 周期间需要进行外周血单个核细胞采集,由陕西医赛尔生物科技有限公司(Shaanxi Yisaier Biotechnology Co., Ltd)完成分选纯化、T 细胞激活、CAR 基因转导、CAR-T 细胞体外扩增,经清洗、制剂、冻存、检测、放行环节后,再以冷链运输到层流病房进行静脉输注。您在接受 CAR-T 细胞治疗前 3-7 天需进行去淋巴化疗重构免疫环境,首选方案为环磷酰胺(CTX)400mg/d,连续两天,第三天检测外周血淋巴细胞清除程度,若清除效果不佳,予以氟达拉滨(Flu)25 mg/m2/d,1~2 天。您在去淋巴化疗后>2 天后,将接受 CD19 CAR-T(1×106/kg)回输,细胞静脉输注前预防性应用抗组胺药物(如氯苯那敏或苯海拉明)和对乙酰氨基酚。随后,您将在层流病房至少住院观察 10 天,若期间您出现 3 级以上细胞因子释放综合征(CRS)等严重不良事件,住院时间将延长至 14 天。整个研究计划随访周期为 1 年,研究结束后的超长期随访将一直进行。

#### 1、入选标准

- (1) 经肾活检确诊为原发性膜性肾病(PMN);
- (2) 中等风险或高风险的难治性膜性肾病;

- (3) 年龄≥18 周岁的患者:
- (4) eGFR≥30 ml/min/1.73m<sup>2</sup>,且无严重心、肝、肺功能异常;
- (5) 签署书面知情同意书。
- 2、排除标准
- (1) 继发性膜性肾病:
- (2)活动性细菌、真菌、病毒(非普通感冒/流感)感染需静脉抗生素治疗,或活动性肺结核,或乙肝病毒(HBV)、丙肝病毒(HCV)、艾滋病毒(HIV)、梅毒螺旋体(TP)、EB病毒(EBV)或巨细胞病毒(CMV)血清学阳性;
  - (3) 严重合并症或基础疾病;
  - (4) 恶性肿瘤史;
  - (5) 治疗史排除,符合下列任意一个条件:
    - a.既往接受过任何细胞治疗(如间充质干细胞等);
  - b.入组前 24 周接受大手术,或计划在入组后 24 周内接受手术;
  - c.计划 3 年内进行肾移植;
  - d.药物滥用史。
  - (6) 入组前3个月内参加过其他干预性临床试验;
  - (7) 妊娠期、哺乳期女性;
  - (8) 无法理解研究或提供知情同意(如严重痴呆、精神疾病);
  - (9) 存在任何研究者认为可能增加风险、干扰评估或影响依从性的情况。
  - 3、终止研究标准

研究受试者的退出标准包括:

- (1) 清除淋巴细胞阶段发生严重不良事件;
- (2) CAR-T 细胞注射时出现严重的不耐受反应;
- (3) 受试者失访、死亡;
- (4) 受试者或其法定监护人自愿提出退出申请;
- (5) 经研究人员评估不宜继续进行试验。

#### 四、研究过程

- 1. 在您入选研究前,医生将询问、记录您的病史,评估患者病情。如符合纳入标准,且您自愿参加研究,将签署知情同意书。如您不愿参加研究,不会导致对您的偏见或影响对您的医疗护理。
  - 2. 若您自愿参加研究,将按以下步骤进行:

若您是合格的纳入者,您可自愿参加研究,签署知情同意书。医师按标准予以 CAR-T 细胞治疗。

主要的干预措施包括:

- (1) 外周血单个核细胞采集。利用血液成分分离机采集您的血液,分离含有 T 细胞的血液。预计采集血量体积为 120ml,最少不低于 50 ml。采集过程中,血液流速设定在 50~70 ml/min,必要时,采集人员将根据实际收集情况调整收集速度,采集时间预计在 2~4 小时。
- (2)淋巴细胞清除化疗。研究将采用环磷酰胺±氟达拉滨方案,经全面评估您的状态,确认您能够耐受淋巴细胞清除化疗后,予以环磷酰胺 400 mg/d,静脉注射,连续两天,总剂量 800 mg,第三天检测外周血淋巴细胞清除程度,若清除效果不佳则可能追加氟达拉滨 25 mg/m²/d,1~2 天。
- (3)自体 CD19 CAR-T 细胞注射液回输。回输前 30~60 分钟使用对乙酰氨基酚衍生物和抗组胺药物(如氯苯那敏或苯海拉明)等。CD19 CAR-T 细胞注射液采用静脉途径回输治疗,使用不带滤网的输血管,以防止有效细胞成分的丢失而降低疗效。回输程序为:生理盐水 100 m1 冲管→细胞回输→生理盐水 100 ml 冲管,前 15min 回输速度控制在 2~3 ml/min,以确保您的耐受性,无不良反应时可改为5~10 ml/min。

同时,在研究期间您需要定期完成随访,主要的随访计划如下:

(1) 密集随访阶段。共计划完成 3 次随访,在接受回输治疗的第 28 天,完成出院后第一次随访(随访 1)。计划完成血尿常规、肝肾功能、凝血功能、C 反应蛋白、降钙素原、抗 PLA2R 抗体、铁蛋白、补体、免疫球蛋白、细胞因子、外周血淋巴细胞亚群、UACR 及 24 小时尿蛋白定量等实验室检查。随后的第二次和第三次随访(随访 2 和 3)分别为治疗后的第 2 和第 3 月,计划完成血尿常规、肝肾功能、抗 PLA2R 抗体、补体、免疫球蛋白、外周血淋巴细胞亚群、外周血 CD19 B 细胞表达、CAR 拷贝参数、UACR 及 24 小时尿蛋白定量等实验室检查。每次随访也应记录伴随用药情况、生命体征等数据。

- (2) 中长期随访阶段。治疗后第 3 个月至第 12 个月间,每 3 个月完成一次随访,共计 3 次随访计划,分别为随访 4 (治疗后第 6 个月)、随访 5 (治疗后第 9 个月)和随访 6 (治疗后第 12 个月),其中随访 6 也是研究结束随访。每次随访计划完成血尿常规、肝肾功能、抗 PLA2R 抗体、补体、免疫球蛋白、CAR 拷贝参数、UACR 及 24 小时尿蛋白定量等实验室检查。随访 4 还需要完成外周血淋巴细胞亚群、外周血 CD19 B 细胞表达检测。每次随访也应记录伴随用药情况、生命体征等数据。
- (3)超长期随访阶段。该随访阶段为研究后随访,不严格设置随访计划,建议患者每3至6月定期自行前往本中心或就近于当地医疗机构完成必要的实验室和影像学检查。研究团队将持续通过电话、短信、微信等形式持续随访患者基本生命体征与病情变化等情况。

此外,在不同的研究阶段需要您配合完成知情同意书签署、病史信息、查体、 心电图/心脏超声、肾脏评估、常规检查、伴随用药记录、终点结局评估等数据信息的采集,这些信息包括但不限于:

- (1)人口学资料。包括姓名、性别、出生年月、民族、文化程度、职业、婚姻状况、现住址、联系方式。
- (2) 伴随用药记录。主要包括降压、调脂、降糖、免疫调节、辅助治疗、疫苗接种等相关药物的使用情况。
  - (3) 生命体征。主要包括心率、血压、体温等。
  - 3. 需要您配合的其他事项

在研究项目进行期间,有可能会出现关于研究方法的新信息。如果出现了新信息,您的研究医生将会及时告知您,并就您是否还愿意继续参与本研究与您进行讨论。如果您决定继续参与研究,您可能被要求签署一份新的知情同意书。随访阶段,医生可能通过电话、门诊随访等方式了解您的情况。

#### 五、风险与不适

如果在研究期间您出现任何不适,或病情发生新的变化,或任何意外情况,不管是否与研究有关,均应及时通知您的医生,他/她将对此做出判断并给予适当的医疗处理。

CAR-T 细胞回输前需要进行淋巴细胞清除预处理(以下简称清淋)为 CAR-T 细胞创造有利的免疫环境,改善其扩增、持久性和临床活性,同时降低抗 CAR 免疫 第 5 页 共 9 页

应答。清淋潜在并发症包括全血细胞减少、免疫抑制、感染、出血性膀胱炎、肝肾损伤等,期间将每天监测您的生命体征,24小时出入量,每1~2天监测全血细胞计数、肝肾功能等。

CAR-T 细胞回输后常见的副作用包括:细胞因子释放综合征(CRS)、免疫效应细胞相关神经毒性综合征(ICANS)、免疫效应细胞相关噬血细胞性淋巴组织细胞增生症样综合征(IEC-HS)、CAR-T 相关出凝血性疾病(CARAC)、免疫效应细胞相关血液毒性(ICAHT)、B 细胞缺乏症/低丙种球蛋白血症、感染、过敏反应和CAR-T 异常增殖等不良反应。

迄今为止,在 CART 细胞治疗自身免疫性疾病患者的临床试验中,严重不良 反应非常少见。未见威胁生命乃至死亡的病例报道,这可能与自身免疫性疾病患者 B 细胞抗原负荷较 B 细胞恶性肿瘤患者要低有关。尽管如此,当前 CAR-T 细胞治疗肾小球肾炎尤其是膜性肾病的临床试验和受试者仍十分有限,安全性数据需要 谨慎解释,对于可能出现的不良反应,本研究参考中国临床肿瘤学会 (CSCO)CAR-T 细胞治疗恶性血液病指南 (2024 年版)和中国嵌合抗原受体 T 细胞治疗难治性神经系统自身免疫性疾病专家共识 (2025 年版),已经制定相应的临床预防和处置预案,并且研究团队也将在临床期间密切关注并评估您可能出现的 CAR-T 细胞治疗相关的剂量限制性毒性与不良反应,予以积极处置。

#### 六、参加研究可能的受益

直接受益:如您参与本项研究,您在使用 CAR-T 治疗后可能改善您的疾病情况(但不保证);同时,您将得到系统观察和治疗随访,使您的疾病情况得到及时的评估,从而最大程度控制疾病的进展,改善疾病转归。

间接受益:我们希望从您参与的本研究中得到的信息在将来能使与您病情相同的病人受益,为优化难治性膜性肾病的治疗和管理,提供新思路、新方案。

#### 七、研究的费用

若您愿意参加本项临床试验,将免除外周血单个核细胞采集、去淋巴化疗、CAR-T治疗、层流病房住院期间产生的全部药品、护理、实验室检查与影像学检查的费用。在 CAR-T 细胞回输后的 12 个月内,因研究而在正常诊疗计划外新增的费用由研究者承担,包括血清铁蛋白、补体、免疫球蛋白、细胞因子、外周血

淋巴细胞亚群、外周血 CD19 B 细胞表达、CAR 拷贝参数的检测费用和随访计划中额外增加的影像学检查,包括心脏彩超、肾脏/肾血管彩超及胸部 CT。

对于难治性膜性肾病患者,即使不参加研究,仍需进行规范的治疗和定时检查才能最大程度保证治疗的有效性。正常诊疗过程中产生的检查费、药费、治疗费等按照住院收费流程自行缴纳。

#### 八、研究的补偿和赔偿

研究期间,医生将尽全力治疗疾病,预防和减少并发症。研究过程与疾病治疗期间均需定期随访,如发生试验相关损害,将由研究者为您购买的临床试验责任险先行赔付,超出的部分由陕西医赛尔生物科技有限公司根据法律法规给予相应的补偿或赔偿。

#### 九、备选疗法

参加这项研究对于该疾病的诊疗不是必须的。对于该项检查还存在其他的方法可供选择,如:其他对症支持治疗。其获益和风险将与具体的治疗方案有关,您可能从中获得相应并发症的控制或缓解,但同时也可能会出现一些治疗常见的毒副反应。您的研究医生会向您介绍具体的检查或治疗方案并解释接受其他检查或治疗方案时会发生哪些好的和坏的情况。他/她会回答您的所有疑问。

#### 十、个人信息保密

本研究中收集到的信息将作为机密保存在医院。为了保护您的身份,在研究 文件中任何关于您的信息都将使用统一格式的编号,而不是使用您的姓名。所收 集和合并的所有受试者信息中,任何可以帮助识别您的身份的信息都将被去除, 保证有关信息不能链接到一个特定的研究受试者。

伦理委员会和管理当局在不违反适用法律和法规所准许的范围内,在不侵犯 受试者隐私的情况下,直接查阅受试者的原始医疗记录以便核查临床试验程序和/ 或数据(申办方不可以查阅),您或您合法代理人在签署知情同意书时即授权这 种查阅。在适用法律和/或法规准许范围内,有关识别您的记录将保密并且不会公 开,本研究的结果可能在医学杂志中发表或出于科学目的进行分享或由申办者用 于产品研究或改进,但您的身份和个人信息在任何时候都将不会被披露。

#### 十一、退出研究

研究过程中研究医生会考虑您利益最大化,如果觉得您不适合再继续进行试验(包括出现疾病复发、发生无法耐受的毒性反应和严重不良事件等),或者申办方/伦理委员会/国家政府部分要求停止,研究医生会向您主动解释原因并中止您的本次研究。您参加本次研究完全自愿,您有权选择不参加本次研究,也有权随时退出而不会因此受到处罚或利益损失,您的后续治疗不会受到任何影响。如果您准备退出研究,请及时告诉您的研究医生,为了您的安全,他将对您进行一次全面检查和处理。研究者得到可能影响您继续参加试验的信息,会及时通报您或您的监护人。

#### 十二、联系人及联系方式

您可随时了解与本研究有关的信息资料和研究进展,若发生与本研究相关的安全性新信息,我们也会及时通知您。如果您有与本研究有关的问题,或您在研究过程中发生了任何不适与损伤,或有关于本项研究参加者权益方面的问题您可以通过(电话号码: 13488317261)与(研究者: 何丽洁 )联系。

#### 十三、伦理委员会联系方式

如果您对参与本研究的权益和健康有任何问题或诉求,您可以联系西京医院 伦理委员会,联系电话: 029-8477179

## 受试者知情同意签字页

我已详细阅读了以上知情同意书,并理解了研究的目的以及参加研究的可能 受益和风险。研究者已将以上医学术语作了明确解释。我有机会提出问题并且所 有问题均得到了通俗易懂的答复。我可以选择不参加本项研究,或在任何时候通 知负责医生后退出,我的任何医疗待遇与权益不会因此而受到影响。如果我需要 其他治疗,或者我没有遵守研究计划,或者发生了与研究相关的损伤,或者有任 何其他原因,负责医生可以终止我继续参与本项研究。

我已阅读了以上知情同意书并获得副本,我的医师也向我作了详尽的说明。我自愿参加本次临床试验。

| 受试者正楷姓名: | 受试者电话: |
|-------------------------------------|------------------------------------|
| 受试者签名: | 日期: |
| (注:受试者无民事行为能力时, 管受试者及其监护人需要签名) | 需监护人签名;受试者为限制民事行为能力时, |
| 监护人正楷姓名: | 与受试者关系: |
| 监护人签名: | 监护人电话: |
| 日期:(年/月/ | (日) |
| 公正见证人签名(如适用): | 日期: |
| (如果受试者或其监护人无阅读能力<br>阅读知情同意书和其他书面材料, | 7时,要求有一位公正见证人签字,公正见证人<br>并见证知情同意。) |
| 我确认已向病人详尽解释了本临 | 苗床试验的有关内容,包括病人可能的获益和 |
| 风险,并解答了患者提出的所有问题 | <b>返。</b> |
| 研究者签名(正楷): | 日期: |
| 研究者电话: | 日期: |